CLINICAL TRIAL: NCT02494297
Title: Drug Utilization Study on the Prescribing Indications for Cyproterone Acetate and Ethinyl Estradiol in 5 European Countries
Brief Title: DUS on the Prescribing Indications for CPA/EE in 5 European Countries
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: ZEG2014_04
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Hirsutism; Androgenetic Alopecia; Severe Anemia; Seborrhea; PCOS
MeSH Terms: conditions — Hirsutism; Alopecia; Anemia; Dermatitis, Seborrheic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cyproterone Acetate and Ethinyl Estradiol: Users of Diane 35 (EE/CPA, BAY86-5264)

SUMMARY:
This study was designed to compile the reasons and specific indications for the prescription of Cyproterone Acetate combined with Ethinyl Estradiol by Health Care Providers. The primary objective of the study was to characterize the prescribing behaviors for Cyproterone Acetate combined with Ethinyl Estradiol in 5 European countries (Austria, Czech Republic, France, the Netherlands, and Spain), including:

* prescription indications for Cyproterone Acetate combined with Ethinyl Estradiol
* use of Cyproterone Acetate combined with Ethinyl Estradiol in accordance with the updated label
* concomitant use of Cyproterone Acetate combined with Ethinyl Estradiol and combined hormonal contraceptives
* second line treatment with Cyproterone Acetate combined with Ethinyl Estradiol for the indication acne

DETAILED DESCRIPTION:
Cyproterone acetate (CPA) 2mg, in combination with ethinyl estradiol (EE) 35mcg, is a medicinal product currently indicated for the treatment of moderate to severe acne in women of reproductive age. Due to the combination with ethinyl estradiol and the dosing, the preparations also act as effective contraceptives.

In 2012, the French health authority conducted a national review of Cyproterone Acetate combined with Ethinyl Estradiol and highlighted serious thromboembolic events and extensive off-label use of these medicines as a contraceptive only. This triggered an Urgent Union Procedure at the beginning of 2013. The European Medicines Agency's Pharmacovigilance Risk Assessment Committee (PRAC) concluded that the benefits of Cyproterone Acetate combined with Ethinyl Estradiol (cyproterone acetate 2mg / ethinyl estradiol 35mcg) outweigh the risks, providing that several measures are taken to minimize the risk of thromboembolism. These medicines should be used solely for the treatment of moderate to severe acne related to androgen sensitivity and/or hirsutism in women of reproductive age. Since Cyproterone Acetate combined with Ethinyl Estradiol acts as a hormonal contraceptive, women should not take these medicines in combination with hormonal contraceptives. As one of the risk minimization measures, the Market Authorization Holders were required to conduct a number of studies including this drug utilization survey.

This study was a multi-national, cross sectional, prospective, non-interventional, drug utilization study conducted in 5 countries. Study participants were recruited by a network of health care professionals. Physicians collected information from study participants based on questionnaires. This was a one-time survey with no follow-up.

Bayer initiated this study and supported it by an unconditional grant to ZEG. Bayer was not actively involved in the study conduct.

Prolongation of recruitment:

At the beginning of May 2016 the recruitment was finished in 4 of the 5 European countries in which the study was conducted (Austria, Czech Republic, The Netherlands, and Spain). At that point in time, only few patients were enrolled in France because of a delayed recruitment start. Therefore, it was agreed to extend the recruitment phase in France until 31st October 2016, in order to ensure that information on the use of Cyproterone Acetate (combined with Ethinyl Estradiol) would be collected from all participating countries.

ELIGIBILITY:
Inclusion Criteria:

* Women who are prescribed Cyproterone Acetate combined with Ethinyl Estradiol during the study period
* Women who are willing to participate in the drug utilization study

Exclusion Criteria:

* Women who are not willing to sign the informed consent
* Women with a language barrier

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who are prescribed Cyproterone Acetate combined with Ethinyl Estradiol during the study period
Sampling Method: Non-Probability Sample
Enrollment: 1597 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, PhD, MD, MSc, MBA, Principal Investigator — Center for Epidemiology and Health Research Berlin
Locations (1):
- Center of Epidemiology and Health Research, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Study Synopsis from Bayer AG — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_BSP_7261&studyid=2078&filename=17194_Study%20Synopsis_CTP.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from March-2015 to 11-May-2016 in Austria, Czech Republic, The Netherlands and Spain; recruitment in France from January-2016 to 31-October-2016, due to late start. Recruitment was conducted by gynecologists, dermatologists and general practitioners.
Groups:
- Cyproterone Acetate and Ethinyl Estradiol: Users of Diane 35 (EE/CPA, BAY86-5264), uncontrolled, single armed drug utilization study
Period: Overall Study
Arm/Group | Cyproterone Acetate and Ethinyl Estradiol
Started (1,698 patients were recruited 101 patients were excluded due to protocol violations.) | 1597
Completed | 1597 (As there was no Follow-Up in this study, participation equals completion)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cyproterone Acetate and Ethinyl Estradiol
Number analyzed (Participants) | 1597
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (7.92)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 200
  18-24 years | 647
  25-34 years | 533
  35-49 years | 203
  >=50 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1597
  Male | 0
Region of Enrollment [Number; unit: participants]
  Austria | 282
  Czech Republic | 563
  France | 108
  Netherlands | 32
  Spain | 612

OUTCOME MEASURES:

1. Primary Outcome: Drug Utilization Pattern of Cyproterone Acetate and Ethinyl Estradiol
Description: Information was obtained from doctors prescribing CPA/EE. Categories in the Outcom Measure Data Table below are based on current disease status.
Time Frame: within 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cyproterone Acetate and Ethinyl Estradiol
Number analyzed (Participants) | 1597
Participants
  Moderate or severe acne (without hirsutism) | 594
  Acne with hirsutism | 128
  Hirsutism without acne | 106
  Other androgenic diseases and contraception | 769

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored in this study, which was a non-interventional observational cross sectional study on drug utilization patterns that exclusively obtained information at the time point of prescription. There were no questions that could generate adverse events (AEs) and no follow-up questionnaires.
Description: Since this was a drug utilization study, exclusively obtaining information at the time of prescription, no adverse events were reported.
Arm/Group | Cyproterone Acetate and Ethinyl Estradiol
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The data cannot indicate a difference in prescribing habits between participating and non-participating physicians. The information about previous treatments of acne is likely to be incomplete because of recall bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes